

Title: NUVISION NAV Statistical Analysis Plan

Statistical Analysis Plan (SAP)

Clinical Evaluation of Intracardiac Ultrasound with the NUVISION™ NAV Ultrasound Catheter.
"NUVISION NAV Study"
(BWI202104)

**Protocol Version: 2.0** 

This document is a confidential communication. The recipient agrees that no unpublished information contained herein will be published or disclosed without prior written approval. This document may be disclosed to the appropriate ethics committees or to duly authorized representatives of the U.S. Food and Drug Administration or other responsible regulatory authorities, under the condition that they are requested to keep it confidential.

SAP Revision: 1.0 SAP Revision Date: 08APR2024

# NUVISION NAV Study Protocol Version: 2.0

The following individuals have reviewed this version of the Statistical Analysis Plan and are in agreement with the content:

## Signature Page

| Study Biostatistician: | | |
|-----------------------------|----------|------|
| (Print) | (Sign) | Date |
| Head of Biostatistics: | | |
| (Print) | (Sign) | Date |
| Franchise Clinical Study Lo | ead: | |
| (Print) | (Sign) | Date |
| Franchise Clinical Platform | ı Lead : | |
| (Print) | (Sign) | Date |

## **Revision History**

| Revision Number | Revision Date<br>(DD/MM/YYYY) | Reasons for Revision |
|-----------------|-------------------------------|----------------------|
| 1.0 | 08/04/2024 | Original document |

Version 1.0 CONFIDENTIAL Page 3 of 12

## List of Acronyms and Abbreviations

| Acronym/Abbreviation | Expanded Term |
|----------------------|---------------------------------|
| AE | Adverse Event |
| AT | Atrial Tachycardia |
| CV | Cardiovascular |
| ICF | Informed Consent Form |
| LA | Left Atrium |
| LAAO | Left Atrial Appendage Occlusion |
| LV | Left Ventricle |
| NYHA | New York Heart Association |
| PAF | Paroxysmal Atrial Fibrillation |
| PP | Per Protocol |
| PsAF | Persistent Atrial Fibrillation |
| PVC | Premature Ventricular Complex |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| TTE | Transthoracic Echocardiography |
| VT | Ventricular Tachycardia |

Version 1.0 CONFIDENTIAL Page 4 of 12

## **Table of Contents**

| 1 | Study Design6 | |
|-----|----------------------------------------------|---|
| 2 | Treatment Assignment6 | |
| 3 | Randomization and Blinding Procedures6 | |
| 4 | Interval Windows6 | |
| 5 | Levels of Significance6 | |
| 6 | Analysis Sets6 | |
| 7 | Sample Size Justification | |
| 8 | Statistical Analysis Methods | |
| 8.1 | General Conventions | |
| 8.2 | Disposition of Study Subjects | |
| 8.3 | Demographic and Baseline Characteristics | |
| 8.4 | Endpoint(s) and Associated Hypotheses | |
| | 8.4.1 Primary Endpoint(s) | |
| | 8.4.2 Secondary Endpoints | |
| | 8.4.3 Additional Endpoints | |
| 8.5 | Analysis of Primary Endpoint(s)9 | |
| 8.6 | Analysis of Secondary Endpoint(s)9 | |
| 8.7 | Analysis of Additional Endpoint(s)1 | 0 |
| 8.8 | Handling of Missing Data | 0 |
| 8.9 | Subgroup Analysis | |
| 9 | Appendix: Tables, Listings and Graphs Shells | 2 |
| 10 | Reference(s) | 2 |

#### 1 Study Design

This study is a prospective, single arm, non-randomized, open-label, multi-center study. Up to 30 subjects will be enrolled.

Subjects meeting the inclusion / exclusion criteria and who sign the informed consent form (ICF) will be enrolled in this study. The clinical investigation is targeting approximately 4 sites in Europe and Israel.

This study will serve to characterize the performance and safety of using the investigational catheter in procedures for subjects in up to five different subgroups (scar-related AT, PsAF, PAF, VT and PVC). Subjects will be treated per investigator's standard of care and followed until 7 days post-procedure.

The primary objective of this study is to assess the performance and safety of using the investigational catheter.

A secondary objective is to gather physician assessment of deployment, maneuverability, navigational features and imaging quality acquired with the investigational catheter.

#### 2 Treatment Assignment

This is a single arm clinical study and all enrolled patients will use the investigational NUVISION™ NAV Ultrasound Catheter (D-1426-01-SI), which is a sterile, single use, disposable, diagnostic ultrasound imaging catheter designed for intracardiac use. It is built around the core design and technology of the existing NUVISION™ Ultrasound Catheter, 10 Fr (D-1423-01-S).

## 3 Randomization and Blinding Procedures

This is a non-randomized, open-label study.

#### 4 Interval Windows

See Section 14.3 of the study protocol.

## 5 Levels of Significance

All data will be summarized by descriptive analyses. No formal hypothesis testing will be performed. All confidence intervals will use the two-sided 95% confidence level unless otherwise stated.

#### 6 Analysis Sets

**Safety Analysis Set**: The Safety Analysis Set will consist of all enrolled subjects who have undergone insertion of the NUVISION™ NAV Ultrasound catheter.

**Per Protocol (PP) Analysis Set**: The PP Analysis Set will include all enrolled subjects who met the study eligibility criteria and in whom assessments were performed with the NUVISION™ NAV Ultrasound catheter.

#### 7 Sample Size Justification

A sample size of 30 subjects will be enrolled to characterize the performance and safety of the Investigational catheter.

The sample size is selected based on previous experience with similar design in first in human assessments of multi-electrode mapping catheters. This study is meant to characterize the catheter's ability to perform safely in various types of arrhythmias. No clinical claims of effectiveness or patient outcomes will be made from this study.

#### 8 Statistical Analysis Methods

#### 8.1 General Conventions

SAS® version 9.4 or higher will be used for all analysis. Standard descriptive summaries for continuous data include the number of observations with data, number of observations with missing data, mean, standard deviation, median, minimum, and maximum values. For categorical data, the count and percentage will be provided. Percentages will be based on the number of subjects without missing data.

#### 8.2 Disposition of Study Subjects

Subject disposition will be summarized and listed for the subject categories defined in protocol section 10.3 for all subjects. Subject disposition will be summarized using categorical summaries. The number and percent of patients who are enrolled in the study, fail inclusion/exclusion criteria, are included in the safety, and perprotocol analysis sets, complete the study, and prematurely discontinue from the study will be presented. Patients who are prematurely discontinued will be summarized by primary reason for discontinuation.

#### 8.3 Demographic and Baseline Characteristics

Demographic variables will include age and sex. Baseline characteristics will include the primary study arrhythmia/procedure and the number of previous ablation procedures. All demographic and baseline characteristics will be summarized using categorical and continuous summaries, as appropriate, for the Safety Analysis Set. A listing of subject demographic and baseline characteristics will be generated.

Medical history will be presented using the Safety Analysis Set.

Cardiovascular (CV) and Thromboembolic/Cerebrovascular medical history will be collected and summarized using categorical summaries. Each subject will be

counted once under each type of CV and/or thromboembolic/cerebrovascular medical history they have experienced.

The number of subjects with TTE performed and those with pericardial effusion will be presented using categorical summaries. The left ventricle ejection fraction and the maximum dimension of pericardial effusion will be presented in continuous summaries.

The number of subjects with an exam performed to assess the presence of thrombus and whether a thrombus is present will be summarized.

Other medical history, including NYHA class, occurrence of diabetes, and history of bleeding will be summarized similarly.

#### 8.4 Endpoint(s) and Associated Hypotheses

#### 8.4.1 **Primary Endpoint(s)**

**Safety**: Occurrence of serious adverse events within 7 days of index procedure related to the NUVISION™ NAV Ultrasound Catheter

**Performance**: Completion of imaging required for the study procedure with the NUVISION™ NAV Ultrasound Catheter without resort to a non-study ultrasound device

#### 8.4.2 **Secondary Endpoints**

Physician assessment of deployment, maneuverability, navigational features and imaging quality acquired with the NUVISION™ NAV Ultrasound Catheter during the study procedures

Occurrence of all other serious adverse events within 7 days of index procedure (not related to the NUVISION™ NAV Ultrasound Catheter)

Occurrence of non-serious adverse events within 7 days of index procedure related to the NUVISION™ NAV Ultrasound Catheter

#### 8.4.3 Additional Endpoints

Additional Procedural data, including:

- Anatomical structures assessed
- Whether imaging for Left Atrium (LA) and Left Ventricle (LV) volume measurements was done
- Total fluoroscopy time
- Total procedure duration

Additional safety data: All non-serious AEs not related to the investigational catheter

#### 8.5 Analysis of Primary Endpoint(s)

Primary Safety Endpoint is defined as the occurrence of serious adverse events related to the Investigational catheter within 7 days of index procedure. An SAE will be counted as related to the investigational catheter if the relationship to a study catheter is anything other than 'Not Related'.

The number of subjects with SAEs related to the investigational catheter will be summarized in the Safety Analysis Set overall and per procedure type (atrial ablation/ventricular ablation) by System Organ Class and Preferred Term and level of relationship. All tables will present summaries both by subject and by event. If a subject has multiple occurrences of an event within a level of summarization, then for the by-subject summaries only a single occurrence will be counted at each level of summarization at the highest level of severity/relationship; for the by-event summary all events will be counted.

All investigational catheter related SAEs will be listed by System Organ Class and Preferred Term, severity, causality (defined as possible, probable or having a causal relationship to the device and/or procedure), anticipation and outcome.

Primary Performance Endpoint is defined as the completion of imaging required for the study procedure with the NUVISION™ NAV Ultrasound Catheter without resort to non-study ultrasound device(s).

The number of subjects who successfully completed the procedure without resort to a non-study ultrasound device will be summarized overall and per procedure type (atrial ablation/ventricular ablation) for the PP Analysis Set.

A listing of the primary performance endpoint will be provided.

#### 8.6 Analysis of Secondary Endpoint(s)

Secondary Safety Endpoints will be analyzed using the Safety Analysis Set:

- All Serious Adverse Events, excluding investigational catheter related SAE, during the 7-day follow-up period.
- All non-serious Adverse Events related to the investigational catheter during the 7day follow-up period

The number of subjects experiencing serious adverse events excluding investigational catheter related SAE and the number of serious adverse events excluding investigational catheter related SAE will be summarized in the Safety Analysis Set overall and per procedure type (atrial ablation/ventricular ablation) using categorical summaries similar to the primary safety endpoint.

The number of subjects experiencing non-serious adverse events related to the investigational catheter and the number of non-serious adverse events related to the investigational catheter will be summarized in the Safety Analysis Set overall and per

procedure type (atrial ablation/ventricular ablation) using categorical summaries similar to the primary safety endpoint.

All SAEs excluding investigational catheter related SAE and all non-serious AEs related to investigational catheter will be listed by System Organ Class and Preferred Term, severity, causality (defined as possible, probable or having a causal relationship to the device and/or procedure), anticipation and outcome.

A listing of device deficiencies including the category and timing of the device deficiency will also be provided. Each deficiency will indicate whether it results in an adverse event.

Physician feedback on deployment, maneuverability, navigational features and imaging quality acquired with the investigational catheter will be analyzed using the PP Analysis Set. A post-procedure survey will be administered. Each question/subquestion will be answered by the physician using a Likert scale of 1 to 7 (1=poor and 7=excellent) and will be summarized. The summary results of each question will be presented overall and per procedure type (atrial ablation/ventricular ablation) using continuous summaries. A by subject listing including all feedback results will be provided.

#### 8.7 Analysis of Additional Endpoint(s)

Additional Procedural Data will be analyzed overall and per procedure type (atrial ablation/ventricular ablation) using the PP Analysis Set and include the following parameters:

- Whether Imaging for Left Atrium (LA) and Left Ventricle (LV) volume measurements was done;
- Total fluoroscopy time;
- Total duration of the procedure.

For each of the above procedural data, the denominator will be the number of subjects where assessments with the study device are performed. Listings will be provided.

Additional safety data, e.g., all non-serious AEs not related to the investigational catheter will be listed by System Organ Class and Preferred Term, severity, causality (defined as possible, probable or having a causal relationship to the device and/or procedure), anticipation and outcome.

#### 8.8 Handling of Missing Data

No missing data will be imputed in this study. All analyses will be performed using observed data.

#### 8.9 **Subgroup Analysis**

Primary and secondary safety endpoints and primary performance endpoint will be further summarized descriptively in the following subgroups:

- 1. Scar-related Atrial Tachycardia
- 2. Persistent Atrial Fibrillation (PsAF)

- Paroxysmal Atrial Fibrillation (PAF)
   Ventricular Tachycardia (VT)
   Premature Ventricular Complex (PVC)

#### 9 Appendix: Tables, Listings and Graphs Shells

Provide, or reference the document that contains the tables, listings and graphs shells. May be replaced with other document (i.e. simulation reports), as appropriate.

#### 10 Reference(s)

- G. Perk, R. M. Lang, M. A. Garcia-Fernandez, J. Lodato, L. Sugeng, J. Lopez, et al., "Use of real time three-dimensional transesophageal echocardiography in intracardiac catheter based interventions," *J Am Soc Echocardiogr*, vol. 22, no. 8, pp. 865-882, Aug 2009.
- F. F. Faletra, G. Pedrazzini, E. Pasotti, S. Muzzarelli, M. C. Dequarti, R. Murzilli, et al., "3D TEE during catheter-based interventions," *JACC Cardiovasc Imaging*, vol. 7, no. 3, pp. 292-308, Mar 2014.
- E. Anter, J. Silverstein, C. M. Tschabrunn, A. Shvilkin, C. I. Haffajee, P. J. Zimetbaum, et al., "Comparison of intracardiac echocardiography and transesophageal echocardiography for imaging of the right and left atrial appendages," *Heart Rhythm*, vol. 11, no. 11, pp. 1890-1897, Nov 2014.
- G. Rigatelli, F. Dell'Avvocata, M. Giordan, N. Viceconte, R. A. Osanna, G. Braggion, et al., "Usefulness of intracardiac echocardiography with a mechanical probe for catheter-based interventions: a 10-year prospective registry," *J Clin Ultrasound*, vol. 42, no. 9, pp. 534-543, Nov-Dec 2014.
- B. A. Medford, N. W. Taggart, A. K. Cabalka, F. Cetta, G. S. Reeder, D. J. Hagler, et al., "Intracardiac echocardiography during atrial septal defect and patent foramen ovale device closure in pediatric and adolescent patients," *J Am Soc Echocardiogr*, vol. 27, no. 9, pp. 984-990, Sep 2014.
- R. Kabra and J. Singh, "Recent trends in imaging for atrial fibrillation ablation," *Indian Pacing Electrophysiol J*, vol. 10, no. 5, pp. 215-227, May 2010
- W. Lee, W. Griffin, D. Wildes, D. Buckley, T. Topka, T. Chodakauskas, et al., "A 10-Fr ultrasound catheter with integrated micromotor for 4-D intracardiac echocardiography," *IEEE Trans Ultrason Ferroelectr Freq Control*, vol. 58, no. 7, pp. 1478-1491, Jul 2011.
- F. E. Silvestry, M. B. Kadakia, J. Willhide and H. C. Herrmann, "Initial experience with a novel real-time three-dimensional intracardiac ultrasound system to guide percutaneous cardiac structural interventions: a phase 1 feasibility study of volume intracardiac echocardiography in the assessment of patients with struc," *J Am Soc Echocardiogr*, vol. 27, no. 9, pp. 978-983, Sep 2014.